CLINICAL TRIAL: NCT04800952
Title: Pharmacokinetics of New Licensed Antibiotics in Critically Ill Patients Receiving Continuous Venovenous Haemofiltration: An International Collaborative Study
Brief Title: Pharmacokinetics of Antibiotics in Critically Ill Patients Receiving CVVHF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Osaka University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20235
Record Dates: First submitted 2021-01-24; First posted 2021-03-16 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Sepsis; Acute Kidney Injury
MeSH Terms: conditions — Sepsis; Acute Kidney Injury | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- To establish the appropriate dosing regimens of newly available antibiotics during CRRT (Other): High dose (world standard dose) and low dose CRRT (Japan local) CRRT protocol Vascular access will be obtained by inserting a double-lumen dialysis catheter into the internal jugular or femoral veins. High dose CRRT in Australia, Blood flow through the extracorporeal circuit will be maintained at 150 ml/min. The CVVHF replacement volume will be set at 25ml/kg/hour and bicarbonate-buffered replacement fluids will be added in post-dilutional mode. Low dose CRRT in Japan, Blood flow through the extracorporeal circuit will be maintained at 80 ml/min. CVVHF replacement volume will be set at 15ml/kg/hour and bicarbonate-buffered replacement fluids will be added in the post-dilutional mode. Fluid balance, volume removal and the duration of CVVHF will be determined by the ICU physician based on the patient's individual clinical status.
  Interventions: Other: blood samples and filtered fluid will be collected.

INTERVENTIONS:
Other: blood samples and filtered fluid will be collected. — Arterial blood samples will be collected just before the commencement of continuous venovenous haemofiltration (CVVHF) and 1 h after the termination of CVVHF.
  Prefilter and post-filter venous blood samples and filtered fluid will be collected 1 and 3 h after the commencement of CVVHF and at the end of CVVHF.

SUMMARY:
The mortality in patients with sepsis and severe acute kidney injury requiring continuous renal replacement therapy (CRRT) remains high. Antibiotic therapy is a key treatment of these patients and in recent years new antibiotics have been licensed. However, data is lacking to determine the optimal dosing regimens of these antibiotics for high (Australia and other countries) and low intensity (Japan) of CRRT.

Aim To establish the appropriate dosing regimens of newly available antibiotics during CRRT can applied globally.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age ≥18 years or older)
* Sepsis (Sepsis-3 criteria)
* Acute kidney injury requiring CRRT (KDIGO criteria)
* Eligible for intensive care without restrictions or limitations

Exclusion Criteria:

* Chronic renal failure
* Obvious or suspected pregnancy
* Intracranial bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Plasma new antibiotics concentration during continuous venovenous haemofiltration (CVVHF) in critically ill patients receiving infusion of these drugs. | 72 hours
  New drugs are Tedizolid, Daptomycin (anti-MRSA), Tazobactam/ Ceftolozane (anti-gram negative), Metronidazole (Anti-anaerobic). Plasma antibiotics concentrations will be measured at 5 time-points and prefilter and postfilter plasma and filtered-fluid antibiotics levels will be measured at 3 time-points during CVVHF.
Calculated clearances of new antibiotics during continuous venovenous haemofiltration (CVVHF) in critically ill patients receiving infusion of these drugs. | 72 hours
  New drugs are Tedizolid, Daptomycin (anti-MRSA), Tazobactam/ Ceftolozane (anti-gram negative), Metronidazole (Anti-anaerobic). Total clearance by CVVHF: (Cltotal) = (Cpre - Cpost / Cpre) × Blood flow (ml/min), Clearance by filtration: (Clfil) = (Clfil / Cpre)× replacement volume (ml/min), Clearance by absorption of the filter: (Clab) = (Cltotal) - (Clfil) (ml/min).

SECONDARY OUTCOMES:
Concentration of serum creatinine | through study completion, an average of 1 year
  Concentration of serum creatinine
length of stay in the hospital | up to 30 days, length of stay in the hospital will be calculated using the earliest of date that the subject is medically ready for discharge when captured, the date of discharge
  length of stay in the hospital
ICU Mortality | at ICU discharge assessed up to 30 days
  Mortality at ICU discharge
Hospital Mortality | at hospital discharge assessed up to 30 days
  Mortality at hospital discharge

IPD SHARING:
Plan to Share IPD: Undecided